CLINICAL TRIAL: NCT05709691
Title: Prevention Program of Innovative Physiotherapy Techniques in People With a Physical Neurological Disease: Oculomotor Therapy and Adapted Yoga
Brief Title: Innovative Physical Therapy Modalities in People With a Neurological Disease: Oculomotor Therapy and Adapted Yoga
Acronym: NeuPhysioLRG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Lidia Ramos Gaspar, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMalagaLR
Record Dates: First submitted 2022-12-15; First posted 2023-02-02 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Nervous System Diseases; Oculomotor; Disorder; Physical Dependence; Physical Inactivity; Treatment Adherence
Keywords: Physical Therapy Modalities; Muscular Stretching Therapy; Oculomotor therapy; Adapted Yoga; Technologies
MeSH Terms: conditions — Nervous System Diseases; Sedentary Behavior; Treatment Adherence and Compliance | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: 128 participants were randomized to follow a physiotherapy online program for 6 weeks. Participants will not know in which group they are, oculomotor therapy will only be used in the experimental group. The results will be measured at the end of the study.
Who Masked: Outcomes Assessor
Masking Description: Participants will not know in which group they are, oculomotor therapy will only be used in the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Oculomotor therapy and adapted yoga.
  Interventions: Other: Oculomotor therapy; Other: Adapted yoga
- Active Comparator (Active Comparator): Adapted yoga.
  Interventions: Other: Adapted yoga

INTERVENTIONS:
Other: Oculomotor therapy — Visual exercise to improve oculomotor behavior.
  Other Names: Visual treatment
  Arms: Experimental
Other: Adapted yoga — Muscular Stretching Therapy, postural control, respiratory physiotherapy.
  Other Names: Yoga

SUMMARY:
Physiotherapy is a discipline which englobe not only the rehabilitation of physical pathologies but also their prevention. That is why this study pretends to upgrade this part of the physical therapy specialty while prove new therapies using innovation technologies in people with any physical neurological disease. The main problem that this study pretends to solve is the necessity of develop new activities to improve quality of life and integration in people with any physical neurological disease.

People with any neurological disease used to present visual problems, pain, fatigue, functional dependence, and a bad quality of life and it appears that exercise habits could improve all these deficiencies. However, how could people with any physical neurological disease participate in an integrated way in nowadays physical activities? The main objective of this study is to prove the effectiveness on visual acuity, quality of life, pain decreasing, functional independence and fatigue of physical therapy modalities in people with any physical neurological disease.

The experiment will take part with 128 participants, divided equally in control and experimental groups. Both are going to receive adapted yoga sessions but only experiment group is going to test oculomotor therapy. Descriptive investigation would take part at the end of the intervention to analyze all results.

DETAILED DESCRIPTION:
Participants will complete several questionnaires at the start and at the end of the study, to quantify the progress. Also, a professional will evaluate the sessions.

Sessions are going to be online and offline, and both will be recorded (with the registered permission of the participants), so they could be analyzed lately.

ELIGIBILITY:
Inclusion Criteria:

* Users equal or over 18 years old.
* To have already signed all the obligatory documents.
* To have a physical neurological disease.
* To have an electronic with internet connection.
* To collaborate on the correct develop of the project.

Exclusion Criteria:

* Serious cognitive or physical damage.
* Doctor disapproval.
* Be unable to understand the indications.
* Be unable to read.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (start point) | Baseline.
  Visual acuity is going to be measured by reading performance, in which users must to read aloud a short text and examiner will count the number of words per second.
Visual acuity (final point) | At study completion, immediately after all the sessions, after 6 weeks.
  Visual acuity is going to be measured by reading performance, in which users must to read aloud a short text and examiner will count the number of words per second.
Search strategy (first session) | Baseline, at first session.
  Using flickering letters that users will explain to examiner, number, type, color and orientation.
Search strategy (through sessions) | Through study completion, an average of 6 weeks.
  Using flickering letters that users will explain to examiner, number, type, color and orientation.
Search strategy (sixth session) | At the final intervention, at 6 weeks.
  Using flickering letters that users will explain to examiner, number, type, color and orientation.
Accomplishment registration | After the intervention, at 6 weeks.
  Examiner will take note of the number of sessions carried out and their full compliance.
Quality accomplishment registration | After the intervention, at 6 weeks.
  Examiner will also take note of the quality of the accomplishment of the sessions: position, breathing and resistance.
The McGill Pain Questionnaire (baseline) | Baseline.
  It is a questionnaire to monitor the pain over time and to determine the effectiveness of the intervention. Total score: 0-45, where 0 means no dolor and 45 means the worse outcome.
The McGill Pain Questionnaire (final) | Immediately after the intervention, at 6 weeks.
  It is a questionnaire to monitor the pain over time and to determine the effectiveness of the intervention. Total score: 0-45, where 0 means no dolor and 45 means the worse outcome.
Modified Fatigue Impact Scale (MFIS) (baseline) | Baseline.
  A questionnaire that serves to register the difference fatigue that users could feel after an exercise therapy program. Total score: 0-84, where 0 means no fatigue and 84 means the worse outcome.
Modified Fatigue Impact Scale (MFIS) (final) | Immediately after the intervention, at 6 weeks.
  A questionnaire that serves to register the difference fatigue that users could feel after an exercise therapy program. Total score: 0-84, where 0 means no fatigue and 84 means the worse outcome.
SF-36 health questionnaire (baseline) | Baseline.
  A questionnaire that allows to quantify the quality of life of users. 36 items are measured. Total score: 0-100, where 0 means the worse score (bad health) and 100 means the better score.
SF-36 health questionnaire (final) | Immediately after the intervention, at 6 weeks.
  A questionnaire that allows to quantify the quality of life of users. 36 items are measured. Total score: 0-100, where 0 means the worse score (bad health) and 100 means the better score.
Functional Independence Measure (FIM) questionnaire (baseline) | Baseline.
  A questionnaire that make possible to register the functional independence. FIM scores range from 1 to 7 (1 = total assist and 7 = complete independence).
Functional Independence Measure (FIM) questionnaire (final) | Immediately after the intervention, at 6 weeks.
  A questionnaire that make possible to register the functional independence. FIM scores range from 1 to 7 (1 = total assist and 7 = complete independence).

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín Valero, PhD, Study Director — Universidad de Málaga
Locations (1):
- Universidad de Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
An average of 2 years.